CLINICAL TRIAL: NCT04748952
Title: The Use of Osseodensification for Ridge Expansion and Dental Implant Placement in Narrow Alveolar Ridges: A Prospective Observational Clinical Study
Brief Title: Ridge Expansion by Osseodensification
Status: Completed | Type: Observational
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Rosol Dawod Salman, Bachelor of Dental Surgery (Master's student), University of Baghdad
Other Study IDs: 19931993
Record Dates: First submitted 2021-01-28; First posted 2021-02-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Horizontal Ridge Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Adult with horizontal bone defect: 30 implants will be placed in osteotomy sites prepared by osseodensification for patients with horizontal bone deficiency based on radiographic findings (CBCT).
  Alveolar ridge width will be measured intraoperatively before and after osteotomy site preparation to assess the amount of ridge expansion. Implant stability will be measured immediately after implant installation and 16 weeks later.
  Interventions: Device: Densah burs

INTERVENTIONS:
Device: Densah burs — Osseodensification is a non-excavating implant site preparation technique. It creates a densified layer of surrounding bone through compaction autografting while simultaneously plastically expanding the bony ridge at the same time facilitating for placement of large diameter implants and also avoiding fenestration and dehiscence defects. The autografting occurs along the entire length of the osteotomy through a hydrodynamic process with the use of irrigation. The result is a consistently cylindrical and densified osteotomy.
  Other Names: Osseodensification

SUMMARY:
A prospective observational clinical study guided by the guidelines of Strengthening the Reporting of Observational Studies in Epidemiology (STORBE) in 2014, that conducted to assess amount of ridge expansion obtained by using Dansah burs with simultaneous implant placement.

DETAILED DESCRIPTION:
In this study, 40 implants will be installed in osteotomy sites prepared by Densah burs (osseodensification preparation technique) for patients with horizontal bone deficiency based on radiographic findings (CBCT).

Alveolar ridge width will be measured intraoperatively before and after osteotomy site preparation to assess the amount of ridge expansion. Implant stability will be measured immediately after implant installation and 16 weeks later.

ELIGIBILITY:
Inclusion criteria

1. Healthy adult patients (≥ 18 years) with American Society of Anesthesiologist physical status classification level I (ASA I), of either gender, having single or multiple missing teeth in the maxilla and/or mandible with alveolar ridge width of 3-6 mm measured at the crest using CBCT.
2. Patients should have ≥ 2 mm of trabecular bone core and ≥ 1/1 trabecular to cortical bone ratio to achieve a predictable expansion according to manufacture instruction in ridge expansion protocol provided by Versah©.
3. Adequate vertical bone height of the alveolar ridge for placement of a minimum length of 8 mm dental implant length based on preoperative OPG or CBCT.
4. Patients who were willing to comply with the study and were available for follow-up visits.

Exclusion Criteria:

- 1. Patients with high bone density (more than 850 HU which corresponds to D1 and D2 according to Misch classification(16)) are not suitable for osseodensification.

2. Patient with severe buccal plate undercut or concavity. 3. Active infection or inflammation in the implant zone. 4. Presence of any uncontrolled systemic diseases. 5. Patients with a history of radiotherapy to the head and neck.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy adults with missing one or more tooth with horizontal alveolar bone defect seeking for dental implant treatment
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Alveolar ridge width | 0 day
  Buccolingual alveolar ridge width measured by using bone caliper at the crest before and after osteotomy preparation to assess amount of expansion obtained

SECONDARY OUTCOMES:
Implant stability | T0= Primary implant stability measured immediately after implant installation , T1 = secondary implant stability measured after 16 weeks
  Implant stability will be measured using resonance frequency analysis (RFA) by Osstell Beacon device.

CONTACTS AND LOCATIONS:
Locations (1):
- College of dentistry, Baghdad, Iraq